CLINICAL TRIAL: NCT04037865
Title: A PHASE 1, NON-RANDOMIZED, OPEN LABEL, MULTIPLE DOSE STUDY TO EVALUATE THE PHARMACOKINETICS, SAFETY AND TOLERABILITY OF PF 06651600 IN PARTICIPANTS WITH RENAL IMPAIRMENT AND IN HEALTHY PARTICIPANTS WITH NORMAL RENAL FUNCTION
Brief Title: A Renal Impairment Study for PF-06651600
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to extensive Covid-19 delay.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B7981020
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — PF-06651600

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PF-06651600 Severe Renal Impairment (Experimental): This arm includes participants with severe renal impairment who will receive oral doses of PF-06651600 50 mg on Day 1 through Day 10
  Interventions: Drug: PF-06651600
- PF-06651600 Normal Renal Function (Experimental): This arm includes participants with normal renal function who will receive oral doses of PF-06651600 50 mg on Day 1 through Day 10
  Interventions: Drug: PF-06651600
- PF-06651600 Moderate Renal Impairment (Experimental): This arm is in Part 2 which will be conducted if decision criterion to proceed to Part 2 is met. This arm includes participants with moderate renal impairment who will receive oral doses of PF-06651600 50 mg on Day 1 through Day 10
  Interventions: Drug: PF-06651600
- PF-06651600 Mild Renal Impairment (Experimental): This arm is in Part 2 which will be conducted if the decision criterion to proceed to Part 2 is met. The arm includes participants with mild renal impairment who will receive oral doses of PF-06651600 50 mg on Day 1 through Day 10.
  Interventions: Drug: PF-06651600

INTERVENTIONS:
Drug: PF-06651600 — PF-06651600 50 mg oral tablets will be administered on Days 1 to 10

SUMMARY:
This is a Phase 1 non-randomized, open-label, parallel cohort study of PF-06651600 in subjects with severe renal impairment and subjects without renal impairment (Part 1) and in subjects with mild and moderate renal impairment (Part 2).

DETAILED DESCRIPTION:
This is a Phase 1 non-randomized, open-label, parallel cohort, multi-site study to investigate the effect of renal impairment on the pharmacokinetics, safety and tolerability of PF-06651600 after multiple oral doses of 50 mg daily. Subjects will be selected and categorized into normal renal function or renal impairment groups based on their estimated glomerular filtration rate. Part 1: A total of approximately 16 subjects will be enrolled; approximately 8 subjects with severe renal impairment and approximately 8 with normal renal function. After statistical evaluation of results from Part 1, Part 2 may be conducted with approximately 8 subjects each with moderate and mild renal impairment. The total duration of participation from Screening visit to Day 11 will be a maximum of 39 days and from Screening visit to Follow-up/Contact Visit will a maximum of 73 days.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of >/= 17.5 to </= 40.0 kg/m2; and a total body weight > 50 kg (110 lb)

Additional inclusion criteria for subjects with renal impairment:

* Meet the following eGFR criteria during the screening period based upon MDRD equation:
* Severe renal impairment: eGFR <30 mL/min but not requiring hemodialysis
* Moderate renal impairment (Part 2 only): eGFR >/=30 mL/min and <60 mL/min
* Mild renal impairment (Part 2 only): eGFR between 60 and 89 mL/min
* Any form of renal impairment except acute nephritic syndrome (subjects with history of previous nephritic syndrome but in remission can be included)
* Stable drug regimen

Exclusion Criteria:

* Females of child-bearing potential must use an accepted, highly effective contraceptive method
* Renal transplant recipients
* Urinary incontinence without catheterization
* Subjects with clinically significant infections within the past 6 months prior to first dose of study drug, evidence of active or chronic infection requiring oral treatment within 4 weeks prior, history of disseminated herpes simplex or recurrent or disseminated herpes zoster
* Subjects with malignancy or with a history of malignancy, with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of skin or cervical carcinoma in situ
* HIV, Hepatitis B, or Hepatitis C infection

Additional exclusion criteria for subjects with renal impairment:

* Subjects requiring hemodialysis and peritoneal dialysis
* Screening BP >/=180 mmHg (systolic) or >/=110 mmHg (diastolic)
* Screening 12-lead ECG demonstrating QTcF >470 msec

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Investigational Drug Services (IDS) University of Miami Hospitals and Clinics, Miami, Florida
  - University of Miami Division of Clinical Pharmacology, Miami, Florida
  - Prism Clinical Research, LLC, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Wojciechowski J, S Purohit V, Huh Y, Banfield C, Nicholas T. Evolution of Ritlecitinib Population Pharmacokinetic Models During Clinical Drug Development. Clin Pharmacokinet. 2023 Dec;62(12):1765-1779. doi: 10.1007/s40262-023-01318-3. Epub 2023 Nov 2. PMID 37917289
- [Derived] Purohit V, Huh Y, Wojciechowski J, Plotka A, Salts S, Antinew J, Dimitrova A, Nicholas T. Leveraging Prior Healthy Participant Pharmacokinetic Data to Evaluate the Impact of Renal and Hepatic Impairment on Ritlecitinib Pharmacokinetics. AAPS J. 2023 Mar 28;25(3):32. doi: 10.1208/s12248-023-00792-8. PMID 36977960
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981020

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated, only participants with severe renal impairment were enrolled. Therefore, in this study, data were collected only for participants with severe renal impairment.
Groups:
- Severe Renal Impairment: Participants with severe renal impairment were included to receive oral PF-06651600 50 mg daily for up to 10 days from Day 1 to Day 10. Stages of renal impairment were based on Kidney Disease Outcomes Quality Initiative Clinical Practice Guidelines for Chronic Kidney Disease.
Period: Overall Study
Arm/Group | Severe Renal Impairment
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants enrolled in the study.
Arm/Group | Severe Renal Impairment
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean | 59.5 (9.78)
Age, Customized [Count of Participants; unit: Participants]
  <18 Years | 0
  18-44 Years | 1
  45-64 Years | 4
  >=65 Years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7
  Black or African American | 1

OUTCOME MEASURES:

1. Primary Outcome: Plasma PF-06651600 Maximum Plasma Concentration (Cmax)
Description: The plasma PF-06651600 Cmax was observed directly from data.
Time Frame: On Day 8 and Day 9 predose, and at 0 (predose), 0.25, 0.5, 1, 2, 4, 6, 8, 12, 16 hours after dose on Day 10, and 24 hours after dose on Day 11.
Population: The analysis population included all participants assigned to investigational product and treated who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Severe Renal Impairment
Number analyzed (Participants) | 8
nanogram per milliliter (ng/mL) | 445.6 (21)

2. Primary Outcome: Plasma PF-06651600 Area Under the Concentration-Time Curve From Time 0 to 24 Hours (AUC0-24)
Description: Plasma PF-06651600 AUC0-24 was determined using a linear/log trapezoidal method.
Time Frame: as for outcome 1
Population: The analysis population included all participants assigned to investigational product and treated who had at least 1 of the PK parameters of primary interest measured.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Severe Renal Impairment
Number analyzed (Participants) | 8
nanogram*hour per milliliter (ng*hr/mL) | 986.3 (33)

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE is considered a TEAE is the event started during the effective duration of treatment. All events that started on or after the first dosing day and time/start time, if collected, but before the last dose plus the lag time were flagged as TEAEs. An AE was considered treatment-related if the causality of the AE was assessed to be the investigational product. The causality of AEs was assessed by the investigator using clinical judgment.
Time Frame: From Screening (Day -28) through and including up to 35 calendar days after the last administration of investigational product, assessed up to 74 days.
Population: The analysis population included all participants assigned to investigational product and who took at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Renal Impairment
Number analyzed (Participants) | 8
Participants
  All-causality TEAEs | 3
  Treatment-related TEAEs | 2

4. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Safety laboratory assessments include clinical chemistry, hematology and urinalysis. Serum creatinine was only assessed on Screening visit 2 and on Day 2 and Day 8 for eGFR assessment. The number of participants with laboratory test abnormalities without regard to baseline abnormality was reported.
Time Frame: At Screening Visit 1 and on Days -1, 5, 11 and early termination day.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Renal Impairment
Number analyzed (Participants) | 8
Participants
  Erythrocytes <0.8xlower limit of normal (LLN) | 1
  Erythrocytes mean corpuscular hemoglobin >1.8*upper limit of normal (ULN) | 1
  Lymphocytes/leukocytes <0.8*LLN | 2
  Eosinophils/leukocytes >1.2*ULN | 1
  Blood urea nitrogen >1.3*ULN | 8
  Creatine >1.3*ULN | 8
  Urate >1.2*ULN | 6
  Bicarbonate <0.9*ULN | 1
  Glucose >1.5*ULN | 1
  Urine glucose >=1 | 2
  Urine protein >=1 | 6
  Urine hemoglobin >=1 | 3
  Leukocyte esterase >=1 | 2

5. Secondary Outcome: Number of Participants With Vital Signs Data Meeting Pre-specified Criteria
Description: Vital signs evaluations included supine blood pressure (BP), pulse rate, and temperature. Criteria for vital signs values included: supine diastolic BP >= 20 mmHg increase from baseline, supine systolic BP >= 30 mmHg increase from baseline, supine diastolic BP >= 20 mmHg decrease from baseline, and supine systolic BP >= 30 mmHg decrease from baseline.
Time Frame: At screening, on Day 1, Day 5, Day 11 and early termination/discontinuation.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Renal Impairment
Number analyzed (Participants) | 8
Participants | 1

6. Secondary Outcome: Number of Participants With Electrocardiogram (ECG) Data Meeting Pre-specified Criteria
Description: ECG criteria included PR, QT, and QTc intervals and QRS complex. Participants with absolute data value meeting the following criteria were reported: aggregate PR interval value >= 300 msec, aggregate QRS duration value >= 140 msec, absolute QTcF interval value >450 msec and <= 480 msec, or >480 msec and <=500 msec, or >500 msec.
Time Frame: At screening, on Day -1, Day 11 and early termination/discontinuation.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Severe Renal Impairment
Number analyzed (Participants) | 8
Participants
  QRS duration value >= 140 msec | 1
  QTcF interval value >450 msec and <=480 msec | 1

ADVERSE EVENTS:
Time Frame: From Screening (Day -28) through and including up to 35 calendar days after the last administration of investigational product, assessed up to 74 days.
Description: Serious adverse events (SAEs) and non-serious AEs were recorded on the CRF. SAEs were also reported on the Clinical Trial (CT) SAE report form to Pfizer Safety within 24 hours of awareness.
Groups:
- Total: All participants.
Arm/Group | Severe Renal Impairment | Total
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Severe Renal Impairment (N=8) | Total (N=8)
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dry eye (Eye disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
Since the study was terminated, the results of this study was not complete and the interpretation of the study results was limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT04037865/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/65/NCT04037865/SAP_001.pdf